CLINICAL TRIAL: NCT03198858
Title: CAPA-VU Trial Catheter Ablation in Paroxymal Atrial Fibrillation Based on UNIVU
Acronym: CAPA-VU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PV4975
Record Dates: First submitted 2016-04-18; First posted 2017-06-26 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation with Carto® 3 System (Other): Ablation with Carto® 3 System
  Interventions: Procedure: Ablation with Carto® 3 System
- Ablation CartoUnivu™ (Other): Ablation CartoUnivu™
  Interventions: Procedure: CartoUnivu™

INTERVENTIONS:
Procedure: CartoUnivu™ — Ablation with Carto® 3 System and image integration module = IIM, CartoUnivu™
  Arms: Ablation CartoUnivu™
Procedure: Ablation with Carto® 3 System — usual Pulmonary vein isolation Ablation with Carto® 3 System only
  Arms: Ablation with Carto® 3 System

SUMMARY:
CartoUnivu™ module easily integrates into the workflow of PVI with the endpoint of unexcitability of the ablation line without prolonging the procedure time. It is associated with a marked reduction in fluoroscopic dose when compared to a conventional 3D-mapping system.

The aim of this prospective randomized study is to evaluate during pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF) whether the use of the IIM is: 1. feasible, 2. can help to reduce fluoroscopy time and burden and 3. has an influence on the procedure duration.

Study design Prospective, randomized controlled multicenter trial, open label. Randomization 1:1

DETAILED DESCRIPTION:
Catheter ablation (CA) has been established as a standard treatment especially in the setting of symptomatic paroxysmal atrial fibrillation (PAF) by means of pulmonary vein isolation (PVI) as recommended in the current guidelines. However, limitations regarding the success rate but also the x-ray burden with regard to patient and operator remain. One of the fundamental disadvantages of CA as it is routinely performed today, based on sequential application of radiofrequency current (RFC), is the need to verify the catheter position throughout the procedure by using fluoroscopy. Catheter guidance in the left atrium has been facilitated by the introduction of three-dimensional mapping systems allowing catheter localization by either weak magnetic or electrical fields with a consecutive reduction of fluoroscopy burden. Nevertheless, despite these 3D mapping systems the fluoroscopy exposure to patient and particularly electrophysiologists is considerable over time. Potential complications associated with radiation exposure include acute and subacute skin injury as well as radiation-induced cancer and genetic abnormalities.

Recently, a new image integration module (IIM, CartoUnivu™ Module) has been introduced allowing the combination and integration of fluoroscopic images within the 3D electroanatomic map. Thus, an accurate navigation without the use of fluoroscopy after acquisition of a left atrial (LA) angiography is possible throughout the procedure. This implies the generation of the 3D left atrial map and catheter navigation for mapping and ablation.

The potential benefit of the new image integration module has been showing the recent pilot study.

The procedural endpoint is the unexcitability of the ablation line after isolation of the pulmonary veins, as described in detail previously. Catheter manipulation should be guided by 3D mapping if safe and feasible to minimize fluoroscopy time in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent
* Symptomatic Paroxysmal Atrial Fibrillation with indication for ablation

Exclusion Criteria:

* Age < 18 years
* Persistent or Permanent Atrial Fibrillation (failed Cardioversion or episode duration > 12 months)
* Previous surgical or interventional therapy of atrial fibrillation
* BMI > 30
* Pregnant women or women of childbearing potential without a negative pregnancy test within 48 hours prior to treatment
* History of hemorrhagic diathesis or other coagulopathies
* Contraindications for oral anticoagulation
* Hyper- or hypothyroidism
* Has any condition that would make participation not be in the best interest of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Radiation duration | 1 year follow up
  Reduction of radiation duration during ablation

SECONDARY OUTCOMES:
procedure duration | 1 year follow up
  Reduction of procedure duration during ablation

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Willems, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Herzzentrum der Universität zu Köln, Cologne
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No